CLINICAL TRIAL: NCT04815174
Title: Observational Study of the Clinico-biological Evolution and Standard of Care Offered to Patients With Ebola Virus Disease
Acronym: EVISTA
Status: Completed | Type: Observational
Sponsor: Alliance for International Medical Action (Other)
Responsible Party: Sponsor
Other Study IDs: ALIMA01
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of Care — (i) advanced clinical and biological monitoring system (ii) symptomatic treatment adapted to the patient's needs, such as antibiotic therapy, oxygen therapy and blood transfusion; (iii) dialysis or mechanical ventilation.

SUMMARY:
This study highlighted the possibility, even in epidemic settings, of providing advanced supportive care for patients with VMEs. Indeed, while the prospect of offering any invasive medical care was widely discussed in 2014 in West Africa with the aim of limiting the exposure of caregivers, the epidemic of 2018-2019 has on the contrary seen the development of a number of medical care strategies, in parallel with the deployment of specific treatments. This study aims to describe a cohort of patients receiving this upgraded supportive care during the tenth epidemic in the DRC.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed Ebola Virus Disease

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with positive RT-PCR admitted in ETC's during the inclusion period were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 711 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Through the end of the hospitalization, with an average of 11 days
  Any type mortality during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- BENI ETC, Beni, North Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided